CLINICAL TRIAL: NCT00003473
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Mixed Glioma
Brief Title: Antineoplaston Therapy in Treating Patients With Recurrent or Refractory Mixed Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066510; BC-BT-18 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Mixed Gliomas
Keywords: recurrent adult mixed glioma; refractoy adult mixed glioma
MeSH Terms: conditions — Glioma | interventions — antineoplaston A10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Atengenal; Drug: Astugenal

INTERVENTIONS:
Drug: Atengenal — Adults with a recurrent or refractory mixed glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10
Drug: Astugenal — Adults with a recurrent or refractory mixed glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: AS2-1

SUMMARY:
RATIONALE: Current therapies for adults with recurrent or refractory mixed gliomas provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with recurrent or refractory mixed gliomas.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with recurrent or refractory mixed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with recurrent or refractory mixed gliomas as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults with recurrent or refractory mixed gliomas.

OVERVIEW: This is a single arm, open-label study in which adults with recurrent or refractory mixed gliomas receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable primary mixed glioma that is recurrent or refractory following standard therapy, including radiation therapy
* Evidence of recurrent or refractory tumor by MRI scan performed within two weeks prior to study entry
* Must have received and failed standard therapy
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/mL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* No renal insufficiency
* Creatinine no greater than 2.5 mg/mL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No known chronic heart failure
* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease
* No severe chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No other severe medical illness
* No nonmalignant systemic disease
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy (unless there is evidence of disease progression)

Surgery:

* Fully recovered from prior surgery

Other:

* Prior cytodifferentiating agent allowed
* No prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1996-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty patients were recruited between March 1996 and May 2008. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal, to mitigate adverse reactions to treatment, until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a recurrent or refractory mixed glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 20
Completed | 17
Not Completed | 3
Not completed — Three patients were not evaluable. | 3

BASELINE CHARACTERISTICS:
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a recurrent or refractory mixed glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: Years] | 37.3 [26.7 to 54.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 17
Participants
  Complete Response | 3
  Partial Response | 0
  Stable Disease | 4
  Progressive Disease | 10

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 20
Percentage of participants
  6 months overall survival | 65.0
  12 months overall survival | 55.0
  24 months overall survival | 30.0
  36 months overall survival | 30.0
  48 months overall survival | 20.0
  60 months overall survival | 15.0

ADVERSE EVENTS:
Time Frame: 10 years, 4 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=20)
Central venous catheter infection (Infections and infestations) | 1 — The central venous catheter infection was not related to Antineoplaton therapy.
Non-functional central venous catheter (General disorders) | 1 — The non-functional venous catheter was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 2 — Neither of the seizures were related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — none of the somnolences/depressed levels of consciousness were related to Antineoplaston therapy.
Pain: Head/headache (Nervous system disorders) | 3 — None of the pain: head/headaches were due to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 1 — The thrombosis/thrombus/embolism was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=20)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Allergy/Immunology - Other (Immune system disorders) | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Hearing (without monitoring program) (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 4
Palpitations (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Central Venous Catheter Infection (Infections and infestations) | 1
Central Venous Catheter Non-functional (General disorders) | 6
Central Venous Catheter Thrombosis/embolism (General disorders) | 1
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13
Fever (General disorders) | 5
Insomnia (General disorders) | 1
Rigors/chills (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 7
Cushingoid appearance (Endocrine disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 9
Hemorrhage, GI: Upper GI NOS (Gastrointestinal disorders) | 1
Hemorrhage, GU (Renal and urinary disorders) | 1
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 3
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1
Infection: Mucosa (Infections and infestations) | 1
Infection: Other (Infections and infestations) | 1
Infection: Stomach (Infections and infestations) | 1
Infection: Upper airway (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2
Hypercholesteremia (Investigations) | 3
Hyperglycemia (Investigations) | 3
Hypernatremia (Investigations) | 15
Hypertriglyceridemia (Investigations) | 2
Hypocalcemia (Investigations) | 1
Hypoglycemia (Investigations) | 6
Hypokalemia (Investigations) | 16
Hypomagnesemia (Investigations) | 1
Hypophosphatemia (Investigations) | 5
Metabolic/Laboratory - Other (Investigations) | 3
Proteinuria (Investigations) | 2
SGOT (Investigations) | 2
SGPT (Investigations) | 4
Uric acid, serum-high (hyperuricemia) (Investigations) | 2
Muscle weakness: Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 5
Confusion (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 2
Mood alteration (Nervous system disorders) | 3
Mood alteration: Agitation (Nervous system disorders) | 1
Neuropathy - cranial (Nervous system disorders) | 1
Neuropathy - motor (Nervous system disorders) | 3
Neuropathy: CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 2
Psychosis (hallucinations/delusions) (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 6
Somnolence/depressed level of consciousness (Nervous system disorders) | 11
Speech impairment (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 3
Diplopia (Eye disorders) | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Vision-photophobia (Eye disorders) | 2
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Pain: Back (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 11
Pain: Joint (Musculoskeletal and connective tissue disorders) | 4
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Pain-Other (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 5
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No